CLINICAL TRIAL: NCT06683404
Title: GISEL (Italian Senologic Group for Electrochemotherapy): Prospective Multicenter Registry of Breast Cancer Patients With Skin Metastases Treated by Electrochemotherapy
Brief Title: GISEL:Registry of Breast Cancer Patients Treated With ECT
Acronym: GISEL
Status: Completed | Type: Observational
Sponsor: Istituto Oncologico Veneto IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: Cod. Int. CE IOV 2017/11
Record Dates: First submitted 2024-01-18; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-01

CONDITIONS: Breast Cancer; Breast Cancer Metastatic; Breast Cancer Recurrent
Keywords: bleomycin; breast cancer; breast cancer cutaneous and subcutaneous metastasis; electrochemotherapy; breast cancer treatment; electroporation
MeSH Terms: conditions — Breast Neoplasms | interventions — Electrochemotherapy; Bleomycin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Breast Cancer patients with cutaneous and/or subcutaneous histologically confirmed metastases: Breast Cancer patients with cutaneous and/or subcutaneous histologically confirmed metastases, regardless of the presence of other metastases, which underwent Electrochemotherapy for the local treatment of their cutaneous and/or subcutaneous metastases.
  Interventions: Device: Electrochemotherapy (ECT); Drug: Bleomycin

INTERVENTIONS:
Device: Electrochemotherapy (ECT) — Electrochemotherapy (ECT) is characterized by the association between the administration of a chemotherapic agent (Bleomycin) with the temporary raise of permeability of the cellular membrane induced by the local administration of electrical impulses (electroporation). ECT represents an effective therapy for loco-regional control of this disease.
Drug: Bleomycin — Electrochemotherapy (ECT) is characterized by the association between the administration of a chemotherapic agent (Bleomycin) with the temporary raise of permeability of the cellular membrane

SUMMARY:
Electrochemotherapy (ECT) is a safe skin-directed treatment for cancer which combines drug treatment with short electric pulses to the tumor. The procedure lasts 20-40 minutes and is generally performed under sedation. It generally allows for a fast recovery with low discomfort.

The aims of this study are to find out how well ECT works in patients with breast cancer that has spread to the skin (cutaneous metastases), and to find out which patients have the best response to the treatment.

DETAILED DESCRIPTION:
In patients with metastatic breast cancer, the skin is affected in 5-30% of cases. Although a relatively uncommon event in absolute terms, the occurrence of skin metastases generally represents an unfavourable prognostic factor (due to simultaneous or imminent disease progression in other sites), as well as a condition of difficult therapeutic management. Even in the most favourable cases, in which the disease is still confined to the locoregional level, cutaneous metastases often entail a worsening of the patients' quality of life, linked to their psychological impact and to the related symptoms (pain, ulceration, bleeding, infection). It is therefore of paramount importance that patients receive timely and effective treatment. Surgical excision represents the simplest and quickest approach to ensure local control of the disease; when the surgical option is not radically feasible, locoregional treatments may be considered. Electrochemotherapy (ECT) has been proposed as a new treatment option for the palliation of skin metastases from breast cancer. Briefly, it consists of the combination of chemotherapy with the local application (at the tumour) of electrical impulses. Through the application of short, intense electrical impulses, a physical phenomenon (reversible electroporation) is produced, which consists of the temporary opening of pores through the cell membrane that increase its permeability. This mechanism allows the diffusion into the cytoplasm of drugs that are in themselves not very permeable. The final effect is an increase in the cytotoxic effect of the drug. The enhancement of cytotoxic action ranges from 80 (in the case of cisplatin) up to 8000 times (in the case of bleomycin). In current clinical practice, ECT is used, as a complementary or alternative treatment, in the management of patients with skin tumours and superficial metastases that cannot be surgically removed or are not amenable to treatment by radiotherapy or systemic oncological therapies. Due to its relative ease of application and favourable toxicity profile, ECT is currently an effective tool for the palliation of symptomatic (bleeding, ulcerated, painful) superficial metastases, thus contributing to the preservation of the patient's quality of life.Recent retrospective studies based on patients with skin metastases from breast cancer treated with ECT found local response rates to treatment of 90%, with 58% of patients reporting complete regression. If these preliminary observations were confirmed in a prospective, larger case series study, the criteria for selecting breast cancer patients eligible for treatment with ECT could be improved.

ELIGIBILITY:
Inclusion Criteria:

1. Cutaneous metastases from breast cancer
2. No indication to surgical resection
3. No indication to treatment with radiotherapy
4. Ineligibility or unresponsiveness to systemic cancer treatment
5. Maximum tumor depth (from the skin layer): 3 cm
6. Patient's life expectancy greater than 4 months
7. Normal hematology, hepatic and renal function
8. Performance status (ECOG) ≤2
9. At least 18 years old

Exclusion Criteria:

1. History of allergic reaction to bleomycin
2. Exceeding the maximum cumulative dose of bleomycin (250,000 IU / m2)
3. Severe impairment of lung, liver or kidney function
4. History of epilepsy
5. Presence of a cardiac pacemaker
6. Serious cardiac arrhythmias
7. Pregnancy or lactation
8. Unwillingness to attend the clinic for follow-up visits
9. Impaired respiratory function or presence of pulmonary fibrosis -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with breast cancer that has spread to the skin (cutaneous metastases), and to find out which patients have the best response to the treatment.
Sampling Method: Probability Sample
Enrollment: 205 (Actual)
Dates: Start 2016-04-22; Primary Completion 2021-10-21 (Actual); Study Completion 2022-12-10 (Actual)

PRIMARY OUTCOMES:
Local response | 4 and 8 weeks
  Local response to the treatment, assessed using clinical examination and graded according to the Response Evaluation Criteria In Solid Tumors (RECIST).
Treatment toxicity | 1 and 2 weeks and 1, 2, 3, 6 and 12 months
  Treatment toxicity, assessed using clinical examination and graded according to the Common Terminology Criteria for Adverse Events (CTCAE v4.0).

SECONDARY OUTCOMES:
Local progression-free survival (LPFS) | 1, 2 , 3 , 6 and 12 months (through study completion, an average of 1 year).
  Local progression-free survival (LPFS), assessed using physical examination
Quality of life and pain relief | 1 and 2 weeks, and at 1, 2, 3, 6 and 12 months
  measured using questionnaire (EQ-5D) EuroQol-5D (The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems) .
Quality of life and pain relief | 1 and 2 weeks, and at 1, 2, 3, 6 and 12 months
  measured using scale (VNS) Verbal Numerical Rating Score (where 0 is no pain and 10 is the worst pain imaginable)

CONTACTS AND LOCATIONS:
Locations (1):
- Veneto Institute of Oncology IRCCS, Padua, Italy

IPD SHARING:
Plan to Share IPD: Yes
The datasets generated during and/or analysed during the current study are/will be available upon request from Prof.Marco Rastrelli (marco.rastrelli@unipd.it)
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Access Criteria: Available on request

REFERENCES:
- [Background] Wong CY, Helm MA, Kalb RE, Helm TN, Zeitouni NC. The presentation, pathology, and current management strategies of cutaneous metastasis. N Am J Med Sci. 2013 Sep;5(9):499-504. doi: 10.4103/1947-2714.118918. PMID 24251266
- [Background] Zagar TM, Higgins KA, Miles EF, Vujaskovic Z, Dewhirst MW, Clough RW, Prosnitz LR, Jones EL. Durable palliation of breast cancer chest wall recurrence with radiation therapy, hyperthermia, and chemotherapy. Radiother Oncol. 2010 Dec;97(3):535-40. doi: 10.1016/j.radonc.2010.10.020. Epub 2010 Nov 11. PMID 21074876
- [Background] Oldenborg S, Van Os RM, Van rij CM, Crezee J, Van de Kamer JB, Rutgers EJ, Geijsen ED, Zum vorde sive vording PJ, Koning CC, Van tienhoven G. Elective re-irradiation and hyperthermia following resection of persistent locoregional recurrent breast cancer: A retrospective study. Int J Hyperthermia. 2010;26(2):136-44. doi: 10.3109/02656730903341340. PMID 20146568
- [Background] Matthiessen LW, Johannesen HH, Hendel HW, Moss T, Kamby C, Gehl J. Electrochemotherapy for large cutaneous recurrence of breast cancer: a phase II clinical trial. Acta Oncol. 2012 Jul;51(6):713-21. doi: 10.3109/0284186X.2012.685524. Epub 2012 Jun 26. PMID 22731832
- [Background] Belehradek M, Domenge C, Luboinski B, Orlowski S, Belehradek J Jr, Mir LM. Electrochemotherapy, a new antitumor treatment. First clinical phase I-II trial. Cancer. 1993 Dec 15;72(12):3694-700. doi: 10.1002/1097-0142(19931215)72:123.0.co;2-2. PMID 7504576
- [Background] Heller R, Jaroszeski MJ, Reintgen DS, Puleo CA, DeConti RC, Gilbert RA, Glass LF. Treatment of cutaneous and subcutaneous tumors with electrochemotherapy using intralesional bleomycin. Cancer. 1998 Jul 1;83(1):148-57. doi: 10.1002/(sici)1097-0142(19980701)83:13.0.co;2-w. PMID 9655305
- [Background] Rodriguez-Cuevas S, Barroso-Bravo S, Almanza-Estrada J, Cristobal-Martinez L, Gonzalez-Rodriguez E. Electrochemotherapy in primary and metastatic skin tumors: phase II trial using intralesional bleomycin. Arch Med Res. 2001 Jul-Aug;32(4):273-6. doi: 10.1016/s0188-4409(01)00278-8. PMID 11440782
- [Background] Mir, LM, Gehl J, Sersa G, et al. Standard operatimg procedures of the electrochemotherapy: instructions for the use of bleomycin or cisplatin administered either systemically or locally and electric pulses delivered by the CliniporatorTM by means of invasive or non-invasive electrodes. Eur J Cancer 2006; 4(suppl 11):14-25
- [Background] Marty M, Sersa G, Garbay JR, et al. Electrochemotherapy - an easy, highly effective and safe treatment of cutaneous and subcutaneous metastases. Results of ESOPE (European Standard Operating Procedures of Electrochemotherapy) study. European Journal of Cancer Supplements 4 (2006) 3-13.
- [Background] Spratt DE, Gordon Spratt EA, Wu S, DeRosa A, Lee NY, Lacouture ME, Barker CA. Efficacy of skin-directed therapy for cutaneous metastases from advanced cancer: a meta-analysis. J Clin Oncol. 2014 Oct 1;32(28):3144-55. doi: 10.1200/JCO.2014.55.4634. Epub 2014 Aug 25. PMID 25154827
- [Background] Cabula C, Campana LG, Grilz G, Galuppo S, Bussone R, De Meo L, Bonadies A, Curatolo P, De Laurentiis M, Renne M, Valpione S, Fabrizio T, Solari N, Guida M, Santoriello A, D'Aiuto M, Agresti R. Electrochemotherapy in the Treatment of Cutaneous Metastases from Breast Cancer: A Multicenter Cohort Analysis. Ann Surg Oncol. 2015 Dec;22 Suppl 3:S442-50. doi: 10.1245/s10434-015-4779-6. Epub 2015 Aug 5. PMID 26242370
- [Background] Campana LG, Valpione S, Falci C, Mocellin S, Basso M, Corti L, Balestrieri N, Marchet A, Rossi CR. The activity and safety of electrochemotherapy in persistent chest wall recurrence from breast cancer after mastectomy: a phase-II study. Breast Cancer Res Treat. 2012 Aug;134(3):1169-78. doi: 10.1007/s10549-012-2095-4. Epub 2012 Jul 24. PMID 22821399
- [Background] Benevento R, Santoriello A, Perna G, Canonico S. Electrochemotherapy of cutaneous metastastes from breast cancer in elderly patients: a preliminary report. BMC Surg. 2012;12 Suppl 1(Suppl 1):S6. doi: 10.1186/1471-2482-12-S1-S6. Epub 2012 Nov 15. PMID 23173816
- [Background] Solari N, Spagnolo F, Ponte E, Quaglia A, Lillini R, Battista M, Queirolo P, Cafiero F. Electrochemotherapy for the management of cutaneous and subcutaneous metastasis: a series of 39 patients treated with palliative intent. J Surg Oncol. 2014 Mar;109(3):270-4. doi: 10.1002/jso.23481. Epub 2013 Oct 28. PMID 24165992
- [Background] Mali B, Jarm T, Snoj M, Sersa G, Miklavcic D. Antitumor effectiveness of electrochemotherapy: a systematic review and meta-analysis. Eur J Surg Oncol. 2013 Jan;39(1):4-16. doi: 10.1016/j.ejso.2012.08.016. Epub 2012 Sep 11. PMID 22980492
- [Background] Therasse P, Arbuck SG, Eisenhauer EA, Wanders J, Kaplan RS, Rubinstein L, Verweij J, Van Glabbeke M, van Oosterom AT, Christian MC, Gwyther SG. New guidelines to evaluate the response to treatment in solid tumors. European Organization for Research and Treatment of Cancer, National Cancer Institute of the United States, National Cancer Institute of Canada. J Natl Cancer Inst. 2000 Feb 2;92(3):205-16. doi: 10.1093/jnci/92.3.205. PMID 10655437
- [Background] Goldhirsch A, Wood WC, Coates AS, Gelber RD, Thurlimann B, Senn HJ; Panel members. Strategies for subtypes--dealing with the diversity of breast cancer: highlights of the St. Gallen International Expert Consensus on the Primary Therapy of Early Breast Cancer 2011. Ann Oncol. 2011 Aug;22(8):1736-47. doi: 10.1093/annonc/mdr304. Epub 2011 Jun 27. PMID 21709140
- [Derived] Russano F, Corrado G, Bonadies A, Migliano E, di Giacomo R, Esposito E, Zamagni C, Ala A, Campana L, Fabrizio T, Ghilli M, Palli D, Renne M, Cabula R, Pelle F, Silvestri B, Dieci MV, Guarneri V, Rastrelli M. Prospective multicentre study of patients with cutaneous metastases from breast cancer treated with electrochemotherapy. Clin Exp Metastasis. 2025 May 29;42(4):32. doi: 10.1007/s10585-025-10350-5. PMID 40439892